CLINICAL TRIAL: NCT05299541
Title: Nutritional Support in Patients Who Have Been Diagnosed at Nutritional Risk in the Hospital and Discharged Home. How we Can Improved the Prognosis and Quality of Life.
Brief Title: Nutritional Support in Patients With Nutritional Risk. How we Can Improved the Prognosis and Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting new subjects
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre Singer, ICU Manager, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0390-16-RMC
Record Dates: First submitted 2022-02-14; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Malnutrition; Quality of Life
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Measurements and questioners
  Interventions: Diagnostic Test: Indirect calorimetric; Diagnostic Test: Bioimpedance; Behavioral: Questioners
- Group A (Active Comparator): Receiving Food dish every night for 6 months Measurements and questioners
  Interventions: Dietary Supplement: Food dish; Diagnostic Test: Indirect calorimetric; Diagnostic Test: Bioimpedance; Behavioral: Questioners
- Group B (Active Comparator): Receiving Food dish every night for 6 months, at this group extra attention have given to the dish plating and appearance by professional (BOCUSE), Measurements and questioners
  Interventions: Diagnostic Test: Indirect calorimetric; Diagnostic Test: Bioimpedance; Behavioral: Questioners; Dietary Supplement: Plated food dish

INTERVENTIONS:
Dietary Supplement: Food dish — All patients will be assessed for nutritional risk estimates (MUST) as well as a nutritional PANDORA estimate that predicts mortality, the Pandora estimate will be measured even after 3 and 6 months
  Group A - will receive a dish of food every evening by a person employed by a rescue organization for 6 months
  At the end of the meal once a week
  * All dishes will be photographed at the end of the meal by Android camera, iPhone
  * A NUTRITION DAY success photo form will be completed and collected .
  Arms: Group A
Diagnostic Test: Indirect calorimetric — • The patient will be measured with an indirect calorimetry device (Fitmate - COSMED Srl. Rome, Italy) to assess the nutritional requirement.
Diagnostic Test: Bioimpedance — • The body composition test will be performed by the Bodystat®4000 Bioimpedance Device (BIA 4000, Bodystat, UK). .
Behavioral: Questioners — At 3 times point , in the recruit + 3 month and 6 month 3 questioners will be given:
  HADS, Quality of life 36SF and FIM
Dietary Supplement: Plated food dish — All patients will be assessed for nutritional risk estimates (MUST) as well as a nutritional PANDORA estimate that predicts mortality, the Pandora estimate will be measured even after 3 and 6 months Group b - will receive a food dish every evening by a person employed by a rescue organization with improved appearance of a plate for 6 months.
  At the end of the meal once a week
  * All dishes will be photographed at the end of the meal by Android camera, iPhone
  * A NUTRITION DAY success photo form will be completed and collected .
  Arms: Group B

SUMMARY:
Background: Many malnourished hospital patients remain after discharge. We aimed to enhance the meal experience after discharge by delivering meals together with physical support at the home and tested if this increased food intake affected survival and quality of life.

Patients and Methods: 60 discharged patients suffering from nutritional (MUST>2) and financial frailty were included. Control group (C) took their regular nutrition at home for 6 months and study group (S) received a daily dinner tray sponsored by the municipality. Hazalla philanthropic organization encouraged the patients at lunch for 6 months. Body composition (Quadstat 4000, Bodystat, UK), energy requirements (Fitmate- COSMED, Italy) were measured at recruitement. Primary outcome was 180 days survival. In addition, in the recruitment stage and after a period of 3 and 6 months, depression and anxiety questionnaire (HADS), quality of Life Questionnaire-SF36and FIM questionnaire - designed to examine the level of independence of patients with disability were performed at days 0, 90 and 180. Statistical analysis used T- Test and ANOVA Repeated Measures. The study was approved by local IRB.

ELIGIBILITY:
Inclusion Criteria:

* MUST =>2
* Region of living Bney-Brak or Petah-tikwa
* Fine cognitive state

Exclusion Criteria:

* Progressive cancer
* Dementia
* Fiddling by PEG or Enteral nutrient via Naso gastric tube
* Psychiatrics disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Improve quality of life | 6 months
  HADS questionnaire (hospital anxiety ans depression scale), scale 0-21. 0-7: normal; 8-10: borderline; 11-21: abnormal.
Improve quality of life | 6 months
  FIM questionnaire (functional indepence measure) scale 0 to 7, 1= total asistance, 7=complete independence, the highst score the best.
Improve quality of life | 6 months
  sf-36 questionnaire (short form health survey), scale 0-100, the highest the score the less disability
changed Mortality | 6 months
  six mounth follow up through ATD (American Trans Data Corp)
changed financials costs per patient in health system | 6 months
  follow up through electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No